CLINICAL TRIAL: NCT02567604
Title: Development of Core Outcomes for Age-related Macular Degeneration (AMD)
Brief Title: Development of Core Outcomes for Age-related Macular Degeneration (AMD) Interventions- Caregivers' Perspective
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Professor Augusto Azuara-Blanco, Professor of Ophthalmology, Queen's University, Belfast
Other Study IDs: B15/31
Record Dates: First submitted 2015-09-11; First posted 2015-10-05 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Focus groups: AMD patients' caregivers defined as people actively taking part in providing support for AMD patients (e.g. family members, unpaid friends, volunteers)
  Interventions: Behavioral: Focus Groups

INTERVENTIONS:
Behavioral: Focus Groups — at least three focus groups lasting approximately one hour
  Other Names: Focus Group Discussion

SUMMARY:
This study will explore experience of AMD caregivers in order to develop a core outcome set (COS) for age related macular degeneration (AMD) randomised controlled trials (RCTs) trying to capture what research outcomes are important from their perspective.

People 18 years of age and older who have been AMD caregivers for at least 6 months may be eligible for this study.

The aim is to conduct three focus groups lasting approximately one hour. The plan is to enrol 18-24 participants (6-8 participants per each of 3 focus groups).Two researchers will be involved in conducting the focus groups. A moderator will ensure fluid discussion, while the second investigator will be taking notes and audio-recording the discussion.

DETAILED DESCRIPTION:
Randomised controlled trials (RCTs) are widely employed interventional studies in medicine, yet many times their outcomes are presented inconsistently. The COMET Initiative (Core Outcome Measures for Effectiveness Trials) suggests that a solution for that issue would be preparation of a core outcome set (COS)a minimal group of outcome measures relevant to different group of stakeholders (e.g. clinicians, patients, carers) that would be implemented in each RCT in a particular area. The overall aim is to prepare a COS for age related-macular degeneration (AMD) RCTs. As first step to develop a COS for AMD, the investigators conducted a systematic review that confirmed variability in AMD trials' outcome selection. The current step encompasses involvement of different stakeholders' groups in focus groups: patients and caregivers (current project) such as family members and friends helping AMD patients with their everyday living. Knowledge of caregivers' perspective on living with, treatment and outcomes for AMD is a key consideration when building up a COS, because they may not only evaluate existing outcomes, but also their experience may be translate into new outcomes. In the current focus group study, caregivers will be invited for a one hour discussion. The investigators plan to arrange three focus groups with approximately 8 participants each. Two researchers will be present to help facilitate discussion. Participants will be asked about their experience related to their help brought to AMD patients, observations of living with and treatment of AMD as well as about AMD study outcomes and their importance.

ELIGIBILITY:
Inclusion Criteria:

* English speaking participants
* AMD patients' caregivers defined as people actively taking part in providing support for AMD patients
* Being a caregiver for at least 6 months
* Having daily contact with AMD patients (not necessarily living with patients)

Exclusion Criteria:

* Non-English speaking participants
* Being a caregiver for less than 6 months
* Not having daily contact with AMD patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: caregivers/ carers such as family members, unpaid friends or volunteers taking active part in providing help and support for AMD patients
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of potential COS (core outcome set) elements for AMD randomised controlled trials as assessed by the focus group discussions. | up to 60 minutes
  The expected list of COS (core outcome set) elements will plausibly include some of the visual function or anatomical measures as well as aspects of the quality of life. This study is a qualitative research study. No interventions will be given to the participants. No questionnaire or scale will be administered. The focus group discussions will aim to explore opinions of caregivers on outcomes used in AMD trials. Repeating themes of the discussions will be captured to form a potential COS for AMD trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Experimental Medicine Queen's University Belfast, Belfast, Co.Antrim, United Kingdom

REFERENCES:
- See also: rationale behind development of core outcome sets for different conditions — http://www.comet-initiative.org/about/overview